CLINICAL TRIAL: NCT00267189
Title: A 6-month, Multicenter, Randomized, Open-label Study of Safety and Efficacy of Everolimus-based Regimen Versus Calcineurin Inhibitor (CNI)-Based Regimen in Maintenance Liver Transplant Recipients
Brief Title: RESCUE Study - Everolimus in Liver Transplantation Recipients With Renal Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001H2401
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation, everolimus, calcineurin inhibitor, renal function
MeSH Terms: interventions — Everolimus; Calcineurin Inhibitors; Cyclosporine; Tacrolimus; Azathioprine; Mycophenolic Acid; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced CNI dose + everolimus ± steroids (Active Comparator): Reduced CNI dose + everolimus (1.5 mg twice daily (b.i.d)) ± steroids
  Interventions: Drug: Everolimus; Drug: Calcineurin inhibitors (CNI); Drug: Steroids
- CNI continuation ± MPA/AZA ± Steroids (Experimental): Standard CNI dose ± MPA/AZA ± steroids
  Interventions: Drug: Calcineurin inhibitors (CNI); Drug: Mycophenolate acid (MPA)/ Azathioprine (AZA); Drug: Steroids

INTERVENTIONS:
Drug: Everolimus — 1.5 mg bid adjusted in order to achieve a trough level between 3 and 8 ng/mL while in combination with CNI and between 6 and 12 ng/mL after CNI discontinuation
  Other Names: Certican; RAD001; Neoral®/Prograf®
  Arms: Reduced CNI dose + everolimus ± steroids
Drug: Calcineurin inhibitors (CNI)
  Other Names: Neoral/Prograf
Drug: Mycophenolate acid (MPA)/ Azathioprine (AZA)
  Other Names: Myfortic/Cellecept
  Arms: CNI continuation ± MPA/AZA ± Steroids
Drug: Steroids

SUMMARY:
The purpose of the study is to assess the effect of everolimus initiation together with reduction or discontinuation of calcineurin inhibitor (CNI) on renal function in maintenance liver transplant recipients with CNI-related renal impairment, while maintaining efficacy.

ELIGIBILITY:
Inclusion criteria

* Male or female 18 - 70 years old
* Patient who has undergone a primary liver transplantation 12 to 60 months ago from a cadaveric or a living donor
* Patient with a calculated GFR ≤ 60 and ≥ 20mL/min
* Patient receiving tacrolimus with C0-h level ≥ 3 and ≤ 8 ng/mL or Neoral® with C0-h level ≥ 50 and ≤ 150 ng/mL or with C2-h level ≥ 250 ng/mL and ≤ 650 ng/mL with or without any of the following (MPA or AZA or steroids)
* Patient willing and capable of giving written informed consent for study participation and able to participate in the study for 6 months
* Patient in whom an allograft biopsy will not be contraindicated
* Female capable of becoming pregnant must have a negative pregnancy test prior to randomization and are required to practice a medically approved method of birth control for the duration of the study

Exclusion criteria

* Recipient of multiple solid organ transplants
* Patient on dialysis
* Patient with an identifiable cause of renal dysfunction other than CNI toxicity
* Patient with proteinuria ≥ 1.0 g/24h
* Patient with any acute rejection within 6 months prior to randomization
* Patient with platelet count of ≤ 50,000/mm³ or white blood cell count of ≤ 2,000/mm³ or hemoglobin value ≤ 8 g/dL
* Undergone a liver transplantation for a hepatocellular carcinoma with sign of recurrence;
* Severe graft dysfunction;
* HCV positive patient who needs an active anti-viral treatment
* HIV positive patient
* Patient who is breast feeding
* Patient with a current severe systemic infection
* Patient who has received an unlicensed drug or therapy within one month prior to study entry
* Presence of any hypersensitivity to drugs similar to everolimus (e.g. macrolides)
* Use of any other immunosuppressive drugs than tacrolimus/cyclosporine microemulsion, steroids, azathioprine and mycophenolic acid

Additional protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigational Site, Germany, Germany
- Novartis Investigative Site, Basel, Switzerland

REFERENCES:
- [Result] De Simone P, Metselaar HJ, Fischer L, Dumortier J, Boudjema K, Hardwigsen J, Rostaing L, De Carlis L, Saliba F, Nevens F. Conversion from a calcineurin inhibitor to everolimus therapy in maintenance liver transplant recipients: a prospective, randomized, multicenter trial. Liver Transpl. 2009 Oct;15(10):1262-9. doi: 10.1002/lt.21827. PMID 19790150
- [Derived] Schrader J, Sterneck M, Klose H, Lohse AW, Nashan B, Fischer L. Everolimus-induced pneumonitis: report of the first case in a liver transplant recipient and review of treatment options. Transpl Int. 2010 Jan;23(1):110-3. doi: 10.1111/j.1432-2277.2009.00900.x. Epub 2009 May 29. No abstract available. PMID 19497063

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Everolimus): Reduced or discontinued CNI dose + everolimus (3-12 ng/mL) ± steroids
- Group 2 (Control): Standard CNI dose ± mycophenolate acid (MPA)/azathioprine (AZA) ± steroids
Period: Overall Study
Arm/Group | Group 1 (Everolimus) | Group 2 (Control)
Started | 72 (Intention to treat (ITT) population.) | 73
Completed Study Medication | 54 | 72
Completed | 67 ("Completed" indicates completed study.) | 72
Not Completed | 5 | 1
Not completed — Patient withdrew consent | 1 | 1
Not completed — Death | 1 | 0
Not completed — Missing | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Everolimus) | Group 2 (Control) | Total
Number analyzed (Participants) | 72 | 73 | 145
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (8.45) | 57.8 (6.93) | 57.4 (7.70)
Age, Customized [Number; unit: Paricipants]
  < 40 years | 1 | 2 | 3
  >= 40 - < 50 years | 12 | 7 | 19
  >= 50 - < 60 years | 29 | 33 | 62
  >= 60 years | 30 | 31 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 60
  Male | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Cockcroft-Gault Calculated Creatinine Clearance (CrCl)
Description: The primary variable was renal function assessed by calculated creatinine clearance using the Cockcroft-Gault formula, and was assessed at all visits.
  CrCl[mL/min] = (140 - A) * W / (72 * C) * R. Where A is age at sample date [years], W is body weight at specific visit [kg], C is the serum concentration of creatinine [mg/dL], R = 1 if the patient is male and = 0.85 if female.
Time Frame: From baseline to 6 months
Population: Intention to treat (ITT) population includes all patients who were randomized to one of the treatment groups and received at least one dose of study medication. Patients with baseline and 6 month creatinine clearance were included in analysis. Missing values at 6 months were imputed using the last observation carried forward (LOCF) approach.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group 1 (Everolimus) | Group 2 (Control)
Number analyzed (Participants) | 71 | 71
mL/min | 0.99 (10.25) | 2.26 (7.79)

2. Secondary Outcome: Percentage of Patients With Efficacy Failure (Biopsy Proven Acute Rejection [BPAR], Graft Loss or Death)
Description: The composite efficacy failure endpoint encompasses at least one of: biopsy proven acute rejection, graft loss, or death for the patient. BPAR was defined as a clinically suspected acute rejection confirmed by biopsy. Acute rejection episodes were recorded as Liver Allograft Rejection. The allograft was presumed to be lost if a patient had a liver retransplant or died.
Time Frame: 6 months
Population: Intention to treat (ITT) population includes all patients who were randomized to one of the treatment groups and received at least one dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | Group 1 (Everolimus) | Group 2 (Control)
Number analyzed (Participants) | 72 | 73
Percentage of patients
  Composite efficacy failure (total) | 2.8 | 1.4
  Biopsy proven acute rejection | 1.4 | 1.4
  Graft Loss | 0 | 0
  Death | 1.4 | 0

3. Secondary Outcome: Number of Patients With Discontinuation of Study Medication
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Group 1 (Everolimus) | Group 2 (Control)
Number analyzed (Participants) | 72 | 73
Patients
  Total # of discontinuation of study medication | 18 | 1
  Adverse Event | 14 | 0
  Patient withdrew consent | 2 | 1
  Abnormal laboratory value(s) | 1 | 0
  Administrative problems | 1 | 0

ADVERSE EVENTS:
Groups:
- Group 1 (Everolimus): Reduced calcineurin inhibitor dose + everolimus (1.5 mg twice daily) ± steroids
- Group 2 (Control): Standard calcineurin inhibitor dose ± mycophenolate acid/azathioprine ± steroids
Arm/Group | Group 1 (Everolimus) | Group 2 (Control)
Serious Adverse Events (participants affected / at risk) | 18/72 | 14/73
Other Adverse Events (participants affected / at risk) | 58/72 | 31/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Everolimus) (N=72) | Group 2 (Control) (N=73)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hyperpyrexia (General disorders) | 2 | 0
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Liver transplant rejection (Immune system disorders) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Everolimus) (N=72) | Group 2 (Control) (N=73)
Anaemia (Blood and lymphatic system disorders) | 6 | 2
Leukopenia (Blood and lymphatic system disorders) | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 11 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Mouth ulceration (Gastrointestinal disorders) | 8 | 0
Nausea (Gastrointestinal disorders) | 6 | 5
Asthenia (General disorders) | 5 | 1
Oedema peripheral (General disorders) | 4 | 1
Pyrexia (General disorders) | 4 | 3
Bronchitis (Infections and infestations) | 4 | 5
Herpes simplex (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 5 | 5
Urinary tract infection (Infections and infestations) | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 4 | 0
Hepatitis C virus (Investigations) | 5 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Headache (Nervous system disorders) | 6 | 2
Renal failure (Renal and urinary disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.